CLINICAL TRIAL: NCT01274481
Title: Effect of Iloprost on Gas Exchange and Pulmonary Mechanics in Patients With Pulmonary Hypertension and ARDS/ALI
Brief Title: Iloprost Effects on Gas Exchange and Pulmonary Mechanics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Actelion (Industry)
Responsible Party: Principal Investigator, Gary Kinasewitz, Principal Investigator, University of Oklahoma
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15123
Record Dates: First submitted 2010-11-15; First posted 2011-01-11 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Lung Injury; Pulmonary Hypertension
Keywords: Acute Respiratory Distress Syndrome; Acute Lung Injury; pulmonary hypertension; oxygenation; lung mechanics; gas exchange
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury; Hypertension, Pulmonary | interventions — Iloprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Iloprost (Experimental): All patients will have their response to Iloprost compared to baseline pre-treatment.
  Interventions: Drug: Iloprost

INTERVENTIONS:
Drug: Iloprost — patients inhale 20 mcg of Iloprost via nebulizer and, if oxygenation and blood pressure is maintained receive a second dose of 20 mcg of Iloprost 30 minutes later.
  Other Names: Ventavis

SUMMARY:
This study will examine the hypothesis that iloprost maintains and improves ventilation perfusion matching in patients with pulmonary hypertension and ARDS/ALI as reflected by 1) an improved PaO2/FIO2 ratio as calculated from the measured arterial blood gases obtained before and after iloprost administration, 2) an improvement in lung compliance, and 3) an improvement in the ventilatory equivalents for oxygen and CO2 measured by expired gas analysis.

DETAILED DESCRIPTION:
Purpose/hypothesis This study will examine the hypothesis that iloprost maintains and improves ventilation perfusion matching in patients with pulmonary hypertension and ARDS/ALI as reflected by 1) an improved PaO2/FIO2 ratio as calculated from the measured arterial blood gases obtained before and after iloprost administration, 2) an improvement in lung compliance, and 3) an improvement in the ventilatory equivalents for oxygen and CO2 measured by expired gas analysis.

Experimental design Twenty patients with pulmonary hypertension and ARDS/ALI will be enrolled. This will be 2-3 hour study conducted on a single day in which each patient's baseline measurements obtained prior to iloprost administration are compared to measurements obtained 30 minutes and 2 hours after Iloprost inhalation. While critically ill by virtue of their underlying illness, patients will be clinically stable over the preceding 2 hours prior to entry into the study as evidenced by airway pressures and arterial O2 saturation that vary less than 10% on the same ventilator settings.

Proposed procedure After baseline measurements are obtained, 10 mcg iloprost will be administered via nebulizer on the inspiratory line of the ventilator. Vital signs including blood pressure and heart rate, respiratory rate and arterial saturation by pulse oximetry will be monitored at baseline and q 5 minutes after the inhalation of iloprost. Thirty (30) minutes after the administration of iloprost the gas exchange, pulmonary function and arterial blood gas measurements will be repeated as described above. Patients who remain clinically stable as evidenced by a fall in arterial PO2 <5 mm Hg, fall in systemic blood pressure of <10% and increase in heart rate of <10 beats/min as well as the absence of symptoms 30 minutes after the inhalation of 20 mcg of iloprost will receive a second dose of 20 mcg. Vital signs will continue to be monitored continuously and 30 minutes after the second dose of iloprost, all pulmonary measurements will be repeated. All patients will be monitored continuously for at least 2 hours after the final dose of iloprost and pulmonary testing will be repeated for a final time 2 hours after the last administration of iloprost. Patients will be deemed to have completed the study after 2 hours provided their vital signs have returned to within 10% of baseline values.

Importance of knowledge reasonably expected to result from the research A positive result in this pilot study will provide a strong rationale leading to a larger long-term study examining the effect of continuous iloprost therapy over several days on pulmonary hemodynamics, gas exchange, and outcome in patients with ARDS/ALI. Markers of inflammation (IL-6 and IL-8), coagulation (thrombin-antithrombin complexes and D-dimer) and collagen formation (TGF* and procollagen peptide III) in lung BAL fluid would be monitored to demonstrate iloprost's potential beneficial effects on lung remodeling in this devastating disorder.

If the research involves more than minimal risk, describe the research plan for monitoring the data collected to ensure the safety of participants.

Data safety monitoring board will meet after the first six patients and determine whether to continue.

ELIGIBILITY:
Inclusion Criteria:

1. Pulmonary hypertension as evidenced by:

   * In patients with a pulmonary artery catheter, a mean pulmonary arterial pressure greater then 25 mmHg with a pulmonary capillary wedge pressure less than or equal to 15 mmHg, or
   * Echocardiographic evidence of pulmonary arterial hypertension including

     * a PA systolic pressure greater than 35 mmHg, or
     * in those patients in whom a PA systolic cannot be estimated for technical reasons, RV dilatation and/or decreased RV function in the presence of normal LV function.
2. ARDS/ALI as indicated by:

   * Diffuse pulmonary infiltrates involving at least three of four quadrants on chest x-ray.
   * PaO2/FIO2 less than 300 while on mechanical ventilation.
   * Recognized cause of ARDS/ALI
   * Absence of clinical evidence of left atrial hypertension
3. presence of an arterial line for pressure monitoring and blood sampling, and
4. the ability to obtain informed consent from the patient or next of kin.

Exclusion Criteria:

1. clinical instability as evidenced by changes in ventilator settings or medications within the preceding hour, and
2. presence of left ventricular dysfunction and/or left atrial enlargement by cardiac echo, or catheterization,
3. Liver failure (Child-Pugh Class B or C)
4. Renal failure on dialysis
5. Pregnancy: all females of child-bearing potential will have a negative pregnancy test before being allowed to enroll
6. Systolic blood pressure less than 85 mm Hg or the need for pressors in the first 10 patients; after review of the first 10 patients by the DMSB, patients on norepinephrine (without additional pressors) in doses less than 0.2 mcg/kg/min may be enrolled if the DMSB finds no evidence of iloprost induced systemic hypotension in the first 10 patients
7. Thrombocytopenia, bleeding diathesis or active bleeding
8. Asthma/Severe bronchospasm
9. Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Arterial oxygenation | 30 minutes

SECONDARY OUTCOMES:
Lung compliance | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gary Kinasewitz, MD, Principal Investigator — University of Oklahoma
Locations (1):
- OU Medical Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Sawheny E, Ellis AL, Kinasewitz GT. Iloprost improves gas exchange in patients with pulmonary hypertension and ARDS. Chest. 2013 Jul;144(1):55-62. doi: 10.1378/chest.12-2296. PMID 23370599